CLINICAL TRIAL: NCT06761456
Title: Development of a Parenteral Injection Training Module and Investigation of Its Effectiveness
Brief Title: Parenteral Injection Training Module
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, lecturer, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17.12.2024-34249
Record Dates: First submitted 2024-12-29; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Injections; Simulation Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working with a training model (Experimental): After the theoretical and skill practice demonstration on parenteral injection application and the application of the pre-test forms, the students were asked to apply parenteral injections using the Clinical Education Module in which 3 Parenteral Interventions could be Applied in the Nursing Fundamentals Laboratory.
  Interventions: Other: Providing training models
- Working without a training model (Active Comparator): After the theoretical and skill practice demonstration on parenteral injection administration and the application of the pre-test forms, the students were asked to apply parenteral injections using a simple model in the Fundamentals of Nursing Laboratory.
  Interventions: Other: Control

INTERVENTIONS:
Other: Providing training models — The experimental group was trained using the Clinical Education Module on 3 Parenteral Interventions in the Nursing Fundamentals laboratory.
  Arms: Working with a training model
Other: Control — The control group was trained using standard training models.
  Arms: Working without a training model

SUMMARY:
Injection practices are a legal obligation of healthcare professionals, but they are also ethically responsible, and the safe maintenance of these practices is extremely important for both patient and employee safety. Due to reasons such as the lack of knowledge and skills of healthcare professionals regarding safe injection, lack of experience, in-service training and periodic training for newly recruited personnel, situations that threaten patient and employee safety occur. Mistakes made in situations requiring technical skills related to injection practices lead to local complications such as ecchymosis, hematoma, pain, abscess, lipodystrophy, infection, and can result in life-threatening situations. In addition, lack of technical skills causes sharp-edge injuries in the world and in excess of their number, and causes blood-borne diseases for many healthcare professionals. In order to prevent these complications and injuries, the education of healthcare professionals requires an education system based on theory and clinical practice, supporting students' cognitive, sensory and psychomotor skills. In the education process, the aim should be to provide clinical skills as well as theoretical knowledge and to develop the acquired skills. Because clinical education allows students to integrate theoretical knowledge with practice in healthcare settings and learn by experience. Gaining competence in parenteral interventions in the clinic is a gradual process and is one of the most important issues in both undergraduate education and postgraduate in-service training. Although clinical practice training is one of the basic practices for learning and acquiring clinical skills in traditional medical and nursing education curricula, it is seen that it is insufficient and it is recommended to benefit from developments in the field of educational technologies in order for practice training to increase patient and student safety. Considering the increasing emphasis on the right of patients to receive care from well-educated health professionals and the right of employees to be safe in risky practices, it is thought that developing a tool that will provide students with the opportunity to practice repeatedly in parenteral injection practice training will be an effective tool in solving all the problems mentioned above. For this purpose, the parenteral practice (intravenous, intramuscular, subcutaneous) skill training module, which is targeted to be developed in the project, aims to improve students' injection skills, provide safe injection practices and ensure their own safety.

ELIGIBILITY:
Inclusion Criteria:

* Students who were 18 years of age or older,
* Enrolled in the Fundamentals of Nursing course,
* Fully participated in the assessments to be applied in the study,
* Volunteered to participate in the study were included in the study

Exclusion Criteria:

* Students who filled in the forms applied within the scope of the study with incomplete information
* Students who dropped out of the Fundamentals of Nursing course while the study was ongoing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Students' self-efficacy scores for applications will increase | 3 weeks
  It is a questionnaire form developed by researchers similar to the Visual Analog Scale (VAS) developed by Hayes and Patterson in 1921, which requires students to evaluate their self-efficacy according to their application skills, with 1 point being the lowest and 10 points being the highest.
The student's satisfaction with the education provided and the self-confidence scale scores in learning will increase. | 3 weeks
  It was developed by Jeffries and Rizzolo (2006) and its Turkish validity and reliability were made by Ünver et al. in 2017 (14). It consists of the subheadings "Satisfaction with Current Learning" and "Self-confidence in Learning". The subheadings of freedom with current learning consist of 5 items, the subheading of diseases in learning consists of 7 items and there are no negative items. It is evaluated that the student's self-confidence in learning has increased. The internal pressure density in temperature is 0.83. Permission to use the scale has been obtained from the author.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol